CLINICAL TRIAL: NCT06970808
Title: Cold SNAre Versus Cold forcePS Polypectomy for Small Colorectal Lesions (Cold-SNAPS): a Multicenter Randomized Trial
Brief Title: Cold Snare Versus Cold Forceps Polypectomy for Small Lesions
Acronym: Cold-SNAPS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda USL Modena (Other)
Responsible Party: Principal Investigator, Dr. Mauro Manno, Gastroenterology and Endoscopy Unit director, Azienda USL Modena
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 04-2025
Record Dates: First submitted 2025-04-27; First posted 2025-05-14 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-04

CONDITIONS: Colorectal Adenoma; Colorectal Lesions
Keywords: Cold forceps polypectomy; Colonoscopy; Cold snare polypectomy

STUDY DESIGN:
Intervention Model Description: Multicenter, Prospective, Randomized, Controlled Study
Masking Description: Only the medical staff who will assess for possible complications, by calling patients 30 days post-polypectomy, will be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cold snare polypectomy group (Active Comparator): For CSP, a 10 mm cold snare will be used (cold snare, Boston Scientific Corporation®, Marlborough, Massachusetts and cold snare, Meditalia S.A.S.®, Palermo, Italy); for CFP, a dedicated forceps will be used (Leviathan® cold forceps, 10 mm opening; Meditalia S.A.S., Palermo, Italy)
  Interventions: Device: Sampling from the resection margins
- Cold forceps polypectomy group (Experimental): For CFP, Leviathan® will be used (Meditalia S.A.S., Palermo, Italy). The opening jaw reaches a 10 mm diameter, and the central section of each jaw has an enlarged diameter up to 3.6 mm compared to the oval axis, enhancing its capacity
  Interventions: Device: Sampling from the resection margins

INTERVENTIONS:
Device: Sampling from the resection margins — After polypectomy, the base will be irrigated and assessed by the endoscopist, who may also use virtual or vital chromoendoscopy, if needed.
  Any residual adenomatous tissue will be removed using the same technique. To confirm the completeness of each polypectomy, two biopsies will be taken from the resection margins for polyps ≤ 5 mm, and three biopsies for polyps 6-9 mm, using standard biopsy forces.

SUMMARY:
The goal of this clinical trial is to compare the efficacy and the safety of a new device for cold forceps polypectomy (CFP)- a special jumbo forceps- to cold snare polypectomy (CSP) for small colorectal lesions, without adding peri- or post-procedural risks to the patient.

The main questions it aims to answer are:

* Does the cold forceps guarantee a complete endoscopic resection rate?
* How many adverse events could the jumbo forceps reduce in comparison to CSP?
* Does the lesion retrieval rate increase?
* Does the polypectomy duration decrease? Participants will be randomized to one or to the other group when a polypoid or non-polypoid lesion is identified. If multiple polyps are found in the same patient, they will be removed using the same polypectomy technique.

If polypectomy cannot be performed using the indicated technique, a crossover will be done according to the best practice of care principles.

DETAILED DESCRIPTION:
The study is a Multicenter, Prospective, Randomized, Controlled Study. It is designed as a non-inferiority trial to assess whether the efficacy in polypectomy of the new jumbo cold forceps is non-inferior to that of the cold snare.

The investigators hypothesize a less number of adverse events with CFP, an increased lesion retrieval rate and a less duration of the polypectomy procedure.

All patients will be contacted, 30 days post-polypectomy, by blinded medical staff assessing for possible complications.

All consecutive patients with polyp lesions can be enrolled, the participation is voluntary and randomization will be performed using the "minimization technique".

ELIGIBILITY:
Inclusion Criteria:

* Patients aged ≥ 18 years;
* Ability to provide informed consent;
* Presence of at least one colorectal polypoid/non-polypoid lesion < 10 mm

Exclusion Criteria:

* Primary or secondary coagulopathy;
* Improper interruption of dual antiplatelet therapy and/or antiplatelet therapy with P2Y12 receptor antagonists (clopidogrel, prasugrel, ticagrelor) and/or anticoagulant therapy;
* Chronic inflammatory bowel diseases;
* Inpatients undergoing colonoscopy;
* Colonoscopy as part of regional colorectal cancer screening;
* Pregnancy or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 312 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2027-10 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Incomplete resection rate | Immediately after the procedure and immediately after the histological evaluation of the biopsy samples
  Compare the rate of incomplete endoscopic resection (IER) of CFP and CSP, defined as the presence of residual adenomatous tissue in the biopsy samples of the margins or after the visual assessment of the resection base.

SECONDARY OUTCOMES:
Adverse events | Up to 30 days after the procedure
  Intraprocedural bleeding (i.e., post-polypectomy "spurting" or "oozing" bleeding lasting more than one minute of observation, requiring hemostatic interventions) and delayed bleeding (within 30 days of the procedure, requiring a second endoscopic treatment and/or hospitalization); perforation (intraprocedural or delayed), defined as grade III (damage to the muscular layer with recognition of the "target sign") or grade IV/V (full-thickness perforation of the bowel wall with or without contamination, respectively) according to the Sydney Classification.
  All patients will be contacted, 30 days post-polypectomy, by blinded medical staff assessing for possible complications (rectal bleeding, abdominal pain, hospitalization due to perforation/bleeding, etc.)
Lesion retrieval rate | During the polypectomy
  Lesion retrieval rate, in relation to the resection site
Polypectomy duration | During the polypectomy
  Polypectomy duration evaluated in seconds: the time will be calculated from the exit of the device from endoscopic channel to the lesion retrieval. Cold forceps polypectomy is assumed to have a shorter procedural time, reducing the overall colonoscopy duration, improving patient compliance, and reducing the sedation required, with fewer risks related to sedation

CONTACTS AND LOCATIONS:
Overall Officials: Mauro Manno, Principal Investigator — AUSL Modena
Locations (1):
- AUSL Modena, Carpi, Modena, Italy

IPD SHARING:
Plan to Share IPD: Undecided